CLINICAL TRIAL: NCT03797326
Title: A Multicenter, Open-label Phase 2 Study of Lenvatinib (E7080/MK-7902) Plus Pembrolizumab (MK-3475) in Previously Treated Subjects With Selected Solid Tumors (LEAP-005)
Brief Title: Efficacy and Safety of Pembrolizumab (MK-3475) Plus Lenvatinib (E7080/MK-7902) in Previously Treated Participants With Select Solid Tumors (MK-7902-005/E7080-G000-224/LEAP-005)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7902-005; MK-7902-005 (Other: MSD Protocol Number); E7080-G000-224 (Other: Eisai Protocol Number); LEAP-005 (Other: MSD); 2018-003747-37 (EudraCT Number)
Record Dates: First submitted 2019-01-07; First posted 2019-01-09 (Actual); Results first posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-10

CONDITIONS: Advanced Solid Tumors; Triple Negative Breast Cancer; Ovarian Cancer; Gastric Cancer; Colorectal Cancer; Glioblastoma; Biliary Tract Cancers; Pancreatic Cancer
Keywords: programmed cell death 1 (PD-1, PD1); programmed cell death ligand 1 (PD-L1, PDL1); programmed cell death ligand 2 (PD-L2, PDL2); tyrosine kinase inhibitor (TKI); multiple TKI; Vascular Endothelial Growth Factor Receptor (VEFG); Fibroblast Growth Factor (FGF); Platelet-Derived Growth Factor (PDGF)
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Ovarian Neoplasms; Stomach Neoplasms; Colorectal Neoplasms; Glioblastoma; Biliary Tract Neoplasms; Pancreatic Neoplasms; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab + Lenvatinib (Arm 1) (Experimental): Participants receive pembrolizumab 200 mg via intravenous (IV) infusion on Day 1 of each 21-day cycle (Q3W) plus lenvatinib 20 mg via oral capsule once a day (QD). Pembrolizumab will be administered for up to 35 cycles (up to 2 years). Lenvatinib will be administered until progressive disease or unacceptable toxicity (up to at least 2 years).
  Interventions: Biological: Pembrolizumab; Drug: Lenvatinib
- Lenvatinib Monotherapy (Arm 2) (Experimental): Participants receive lenvatinib 24 mg via oral capsule QD, to be administered until progressive disease or unacceptable toxicity (up to at least 2 years).
  Interventions: Drug: Lenvatinib

INTERVENTIONS:
Biological: Pembrolizumab — Administered as an IV infusion on Day 1 Q3W.
  Other Names: MK-3475; Keytruda®
  Arms: Pembrolizumab + Lenvatinib (Arm 1)
Drug: Lenvatinib — Administered orally once a day during each 21-day cycle.
  Other Names: MK-7902; E7080; LENVIMA™

SUMMARY:
The purpose of this study is to determine the safety and efficacy of combination therapy with pembrolizumab (MK-3475) and lenvatinib (E7080/MK-7902) in participants with triple negative breast cancer (TNBC), ovarian cancer, gastric cancer, colorectal cancer (CRC), glioblastoma (GBM), biliary tract cancers (BTC), or pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Has a histologically or cytologically-documented, advanced (metastatic and/or unresectable) solid tumor that is incurable and for which prior standard systemic therapy has failed in one of the following cohorts: TNBC, Ovarian Cancer, Gastric Cancer, Colorectal Cancer, GBM, BTC (intrahepatic, extrahepatic cholangiocarcinoma and gall bladder cancer; excludes Ampulla of Vater), Pancreatic Cancer
* Must have progressed on or since the last treatment
* Has measurable disease per RECIST 1.1 (RANO for the GBM cohort) as assessed by the local site investigator/radiology and confirmed by BICR
* Has provided a PD-L1 evaluable archival tumor tissue sample or newly obtained core or excisional biopsy of a tumor lesion not previously irradiated
* Male participants agree to use approved contraception during the treatment period for at least 7 days after the last dose of lenvatinib, or refrain from heterosexual intercourse during this period
* Female participants are not pregnant or breastfeeding, and are not a woman of childbearing potential (WOCBP), OR are a WOCBP that agrees to use contraception during the treatment period (or 14 days prior to the initiation of study treatment for oral contraception) and for at least 120 days post pembrolizumab, or 30 days post lenvatinib, whichever occurs last
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1 within 3 days of study treatment initiation
* Has adequate organ function

For Triple Negative Breast Cancer Participants:

* Has received one or 2 prior lines of therapy
* Has Lactate Dehydrogenase (LDH) <2.0 x Upper Limit of Normal (ULN)
* Has locally determined results for estrogen receptor, progesterone receptor, and human epidermal growth factor receptor 2 tumor analyses

For Ovarian Cancer Participants:

- Has primary ovarian cancer and has received 3 prior lines of therapy.

For Gastric Cancer Participants:

- Has received 2 prior lines of therapy. Note: Gastric cancer will include participants with both gastric and gastroesophageal junction (GEJ) adenocarcinoma. Participants with squamous cell carcinoma histology are not eligible

For Colorectal Cancer Participants:

- Has received 2 prior lines of therapy

For GBM Participants:

* Has failed initial systemic therapy for newly diagnosed GBM
* Have the following time periods elapsed before the projected start of scheduled study treatment: 1) at least 3 weeks from prior surgical resection, 2) at least 1 week from stereotactic biopsy, 3) at least 6 months from completion of prior radiotherapy, 4) at least 4 weeks (or 5 half-lives, whichever is shorter) from any investigational agent, 5) at least 4 weeks from cytotoxic therapy, 6) at least 6 weeks from antibodies, 7) at least 4 weeks (or 5 half-lives, whichever is shorter) from other antitumor therapies and 1 week for cancer vaccines
* Be neurologically stable (e.g. without a progression of neurologic symptoms or requiring escalating doses of systemic steroid therapy within last 2 weeks) and clinically stable
* Has histologically confirmed World Health Organization (WHO) Grade IV GBM
* Has locally determined result for O^6-methylguanine-DNA methyltransferase (MGMT) analysis

For Biliary Tract Cancer Participants:

* Has received 1 prior line of therapy
* Child-Pugh Score, Class A: well-compensated disease. Child-Pugh Score of 5-6

For Pancreatic Cancer Participants:

* Has pathologically (histologically or cytologically) confirmed pancreatic ductal adenocarcinoma that is metastatic at enrollment
* Has received one or 2 prior lines of therapy
* Has received prior therapy with at least 1 (platinum-containing regimen or gemcitabine-containing regimen) but no more than 2 prior systemic therapies for unresectable or metastatic pancreatic cancer

Exclusion Criteria:

* Has gastrointestinal malabsorption or any other condition that might affect the absorption of lenvatinib
* Has present or progressive accumulation of pleural, ascitic, or pericardial fluid requiring drainage or diuretic drugs within 2 weeks prior to enrollment (applies to all cohorts except the ovarian cancer cohort)
* Has radiographic evidence of encasement or invasion of a major blood vessel or of intratumoral cavitation. Participants with portal vein invasion (Vp4), inferior vena cava, or cardiac involvement based on imaging in the BTC cohort are not eligible for enrollment
* Has clinical significant hemoptysis or tumor bleeding within 2 weeks prior to the first dose of study treatment
* Has significant cardiovascular impairment within 12 months of the first dose of study treatment, such as history of congestive heart failure greater than New York Heart Association (NYHA) Class II, unstable angina, myocardial infarction or cerebrovascular accident (CVA), or cardiac arrhythmia associated with hemodynamic instability
* Has a history of arterial thromboembolism within 12 months of start of study treatment
* Has a known additional malignancy that is progressing or has required active treatment within the past 3 years.
* Has a serious nonhealing wound, ulcer or bone fracture
* Has had major surgery within 3 weeks prior to first dose of study interventions
* Has biologic response modifiers therapy (e.g. granulocyte colony-stimulating factor) within 4 weeks before study entry
* Has preexisting ≥Grade 3 gastrointestinal (GI) or non-gastrointestinal fistula
* Has received prior therapy with lenvatinib, an anti-PD-1, anti-PD-L1, or anti PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g. cytotoxic T-lymphocyte-associated protein 4 [CTLA-4], Tumor necrosis factor receptor superfamily, member 4 [OX 40], tumor necrosis factor receptor superfamily member 9 [CD137])
* Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks prior to study treatment start
* If participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment
* Has received prior radiotherapy within 2 weeks of start of study treatment. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-central nervous system (CNS) disease
* Has received a live vaccine within 30 days prior to the first dose of study treatment
* Has known intolerance to lenvatinib (and/or any of the excipients)
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior the first dose of study treatment
* Has known active CNS metastases and/or carcinomatous meningitis
* Has tumors involving the brain stem
* Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients
* Has an active autoimmune disease that has required systemic treatment in past 2 years
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis
* Has an active infection requiring systemic therapy
* Has a known history of human immunodeficiency virus (HIV) infection
* Has a known history of hepatitis B or known active hepatitis C virus infection
* Has a known history of active tuberculosis (TB; Bacillus tuberculosis)
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of study treatment
* Has had an allogenic tissue/solid organ transplant (large organ transplants, stem-cell transplant requiring chronic immunosuppressant therapy necessary to prevent graft rejection)

For GBM Participants:

* Has carcinomatous meningitis
* Has recurrent tumor greater than 6 cm in maximum diameter
* Has tumor primarily localized to the brainstem or spinal cord
* Has presence of multifocal tumor, diffuse leptomeningeal or extracranial disease
* Has evidence of intratumoral or peritumoral hemorrhage on baseline magnetic resonance imaging (MRI) scan other than those that are grade ≤ 1 and either post-operative or stable on at least 2 consecutive MRI scans
* Has received Optune® TTFields within 2 weeks of study intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 611 (Actual)
Dates: Start 2019-02-12 (Actual); Primary Completion 2024-10-28 (Actual); Study Completion 2024-10-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (88):
- United States (14):
  - City of Hope ( Site 0002), Duarte, California
  - Cedars Sinai Medical Center ( Site 0003), Los Angeles, California
  - University of California Davis Comprehensive Cancer Center ( Site 0005), Sacramento, California
  - University of Colorado, Anschutz Cancer Pavilion ( Site 0007), Aurora, Colorado
  - University of Florida-Health Cancer Center-Orlando ( Site 0015), Orlando, Florida
  - Rutgers Cancer Institute of New Jersey ( Site 0009), New Brunswick, New Jersey
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone Health ( Site 0023), New York, New York
  - Sanford Fargo Medical Center ( Site 0059), Fargo, North Dakota
  - Lehigh Valley Hospital- Cedar Crest ( Site 0047), Allentown, Pennsylvania
  - Sanford Cancer Center ( Site 0058), Sioux Falls, South Dakota
  - West Cancer Center - East Campus ( Site 0018), Germantown, Tennessee
  - Mary Crowley Cancer Research Centers - Medical City Hospital ( Site 0049), Dallas, Texas
  - Swedish Medical Center ( Site 0021), Seattle, Washington
  - University of Wisconsin Carbone Cancer Center ( Site 0017), Madison, Wisconsin
- Argentina (6):
  - Fundacion Favaloro para la Docencia e Investigacion Medica ( Site 2106), Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Hospital Aleman ( Site 2100), Buenos Aires, Buenos Aires F.D.
  - Hospital Britanico de Buenos Aires ( Site 2109), Ciudad de Buenos Aires, Buenos Aires F.D.
  - Instituto de Oncologia de Rosario ( Site 2105), Rosario, Santa Fe Province
  - CEMIC ( Site 2104), Buenos Aires
  - IDIM Instituto de Diagnostico e Investigaciones Metabolicas ( Site 2101), Caba
- Australia (3):
  - Royal Brisbane and Women s Hospital ( Site 0901), Herston, Queensland
  - Alfred Health ( Site 0902), Melbourne, Victoria
  - Sir Charles Gairdner Hospital ( Site 0903), Nedlands, Western Australia
- Canada (7):
  - BC Cancer - Abbotsford ( Site 0200), Abbotsford, British Columbia
  - CancerCare Manitoba ( Site 0201), Winnipeg, Manitoba
  - Hamilton Health Sciences-Juravinski Cancer Centre ( Site 0208), Hamilton, Ontario
  - Sunnybrook Research Institute ( Site 0207), Toronto, Ontario
  - Princess Margaret Cancer Centre ( Site 0202), Toronto, Ontario
  - Centre Hospitalier de l Universite de Montreal - CHUM ( Site 0210), Montreal, Quebec
  - CHU de Quebec Universite de Laval ( Site 0206), Québec, Quebec
- Chile (4):
  - Fundacion Arturo Lopez Perez ( Site 1201), Santiago, Region M. de Santiago
  - Pontificia Universidad Catolica de Chile ( Site 1202), Santiago, Region M. de Santiago
  - Hospital Clinico Universidad de Chile ( Site 1200), Santiago, Region M. de Santiago
  - Centro Investigación del Cáncer James Lind ( Site 1203), Temuco, Región de la Araucanía
- Colombia (4):
  - Fundacion Colombiana de Cancerologia Clinica Vida ( Site 1105), Medellín, Antioquia
  - Instituto Nacional de Cancerologia E.S.E ( Site 1102), Bogotá, Bogota D.C.
  - Oncologos del Occidente S.A. ( Site 1106), Pereira, Risaralda Department
  - Fundacion Valle del Lili ( Site 1101), Cali, Valle del Cauca Department
- France (6):
  - Centre Antoine Lacassagne ( Site 0404), Nice, Alpes-Maritimes
  - Centre Leon Berard ( Site 0405), Lyon, Auvergne
  - Institut Claudius Regaud IUCT Oncopole ( Site 0403), Toulouse, Haute-Garonne
  - Centre Oscar Lambret ( Site 0401), Lille, Nord
  - Institut de Cancerologie de l Ouest Centre Rene Gauducheau ( Site 0402), Saint-Herblain, Val-de-Marne
  - Institut Gustave Roussy ( Site 0400), Villejuif, Val-de-Marne
- Germany (6):
  - Robert Bosch GmbH ( Site 0307), Stuttgart, Baden-Wurttemberg
  - Universitaetsklinikum Regensburg ( Site 0304), Regensburg, Bavaria
  - Universitaetsklinikum Frankfurt ( Site 0306), Frankfurt am Main, Hesse
  - HELIOS Dr. Horst Schmidt Kliniken Wiesbaden ( Site 0301), Wiesbaden, Hesse
  - SRH Wald-Klinikum Gera GmbH ( Site 0309), Gera, Thuringia
  - Universitaetsklinikum Jena ( Site 0302), Jena, Thuringia
- Israel (5):
  - Soroka Medical Center ( Site 0601), Beersheba
  - Rambam Medical Center ( Site 0602), Haifa
  - Hadassah Ein Kerem Medical Center ( Site 0604), Jerusalem
  - Chaim Sheba Medical Center ( Site 0600), Ramat Gan
  - Sourasky Medical Center ( Site 0603), Tel Aviv
- Italy (4):
  - Istituto Clinico Humanitas Research Hospital ( Site 1402), Rozzano, Milano
  - Policlinico Le Scotte - A.O. Senese ( Site 1401), Siena, Tuscany
  - Istituto Nazionale Tumori Fondazione Pascale ( Site 1400), Napoli
  - Fondazione Policlinico Universitario A. Gemelli ( Site 1403), Roma
- Russia (6):
  - Arkhangelsk Clinical Oncological Dispensary ( Site 1600), Arkhangelsk, Arkhangelskaya oblast
  - Russian Oncological Research Center n.a. N.N. Blokhin ( Site 1604), Moscow, Moscow
  - Leningrad Regional Oncology Center ( Site 1609), Saint Petersburg, Sankt-Peterburg
  - Scientific Research Oncology Institute n.a. N.N.Petrov ( Site 1610), Saint Petersburg, Sankt-Peterburg
  - City Clinical Oncology Center ( Site 1608), Saint Petersburg, Sankt-Peterburg
  - Republican Clinical Oncology Dispensary of Tatarstan MoH ( Site 1603), Kazan', Tatarstan, Respublika
- South Korea (3):
  - Asan Medical Center ( Site 1002), Songpagu, Seoul
  - Seoul National University Hospital ( Site 1000), Seoul
  - Severance Hospital Yonsei University Health System ( Site 1001), Seoul
- Spain (4):
  - Hospital Clinic i Provincial ( Site 0703), Barcelona
  - Hospital Universitario Gregorio Maranon ( Site 0701), Madrid
  - Clinica Universitaria de Navarra ( Site 0704), Madrid
  - Hospital Ramon y Cajal ( Site 0702), Madrid
- Switzerland (6):
  - Inselspital Universitaetsspital Bern ( Site 1705), Bern, Canton of Bern
  - Kantonsspital St. Gallen ( Site 1702), Sankt Gallen, Canton of St. Gallen
  - Ospedale Regionale di Bellinzona e Valli ( Site 1703), Bellinzona, Canton Ticino
  - Kantonsspital Graubuenden ( Site 1704), Chur, Kanton Graubünden
  - Hopitaux Universitaires de Geneve HUG ( Site 1701), Geneva
  - Universitaetsspital Zurich ( Site 1700), Zurich
- Taiwan (2):
  - National Cheng Kung University Hospital ( Site 3003), Tainan
  - National Taiwan University Hospital ( Site 3000), Taipei
- Thailand (3):
  - Chulalongkorn University ( Site 5001), Bangkok, Bangkok
  - Ramathibodi Hospital. ( Site 5002), Bangkok, Bangkok
  - Siriraj Hospital ( Site 5003), Bangkok, Bangkok
- United Kingdom (5):
  - Cambridge University Hospitals NHS Trust ( Site 0803), Cambridge, Cambridgeshire
  - Leicester Royal Infirmary. Univ. Hosp. of Leicester NHS Trust ( Site 0804), Leicester, Leicestershire
  - Guy's Hospital ( Site 0806), London, London, City of
  - Royal Marsden Hospital (Sutton) ( Site 0800), London, Surrey
  - Christie NHS Foundation Trust ( Site 0805), Manchester

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Gonzalez-Martin A, Chung HC, Saada-Bouzid E, Yanez E, Senellart H, Cassier PA, Basu B, Corr BR, Girda E, Dutcus C, Okpara CE, Ghori R, Jin F, Groisberg R, Lwin Z. Lenvatinib plus pembrolizumab for patients with previously treated advanced ovarian cancer: Results from the phase 2 multicohort LEAP-005 study. Gynecol Oncol. 2024 Jul;186:182-190. doi: 10.1016/j.ygyno.2024.04.011. Epub 2024 May 7. PMID 38718741
- [Result] Chung HC, Saada-Bouzid E, Longo F, Yanez E, Im SA, Castanon E, Desautels DN, Graham DM, Garcia-Corbacho J, Lopez J, Dutcus C, Okpara CE, Ghori R, Jin F, Groisberg R, Korakis I. Lenvatinib plus pembrolizumab for patients with previously treated, advanced, triple-negative breast cancer: Results from the triple-negative breast cancer cohort of the phase 2 LEAP-005 Study. Cancer. 2024 Oct 1;130(19):3278-3288. doi: 10.1002/cncr.35387. Epub 2024 Jun 21. PMID 39031824
- [Derived] Rha SY, Castanon E, Gill S, Senellart H, Lopez J, Marquez-Rodas I, Victoria I, Kim TM, Lwin Z, Burger MC, Simonelli M, Cassier PA, Hendifar AE, Ascierto PA, Dutcus C, Okpara CE, Ghori R, Jin F, Groisberg R, Villanueva L. Lenvatinib plus pembrolizumab for patients with previously treated select solid tumors: Results from the phase 2 LEAP-005 study recurrent glioblastoma cohort. Cancer. 2025 Aug 15;131(16):e70015. doi: 10.1002/cncr.70015. PMID 40808295
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 85 centers in 17 countries.
Groups:
- Cohort A: Triple Negative Breast Cancer (Lenva + Pembro): Participants received Pembrolizumab (pembro) 200 mg via intravenous (IV) infusion on Day 1 of each 21-day cycle (Q3W) for up to 35 cycles (up to 2 years) PLUS Lenvatinib (lenva) 20 mg via oral capsule once a day (QD) up to at least 2 years. Participants continued study intervention until progressive disease or unacceptable toxicity.
- Cohort B: Ovarian Cancer (Lenva + Pembro); Cohort C: Gastric Cancer (Lenva + Pembro); Cohort D1: Colorectal Cancer (Lenva + Pembro); Cohort E: Glioblastoma Multiforma (Lenva + Pembro); Cohort F: Biliary Tract Cancer (Lenva + Pembro); Cohort G: Pancreatic Cancer (Lenva + Pembro): Participants received Pembro 200 mg via IV infusion on Day 1 of each 21-day cycle (Q3W) for up to 35 cycles (up to 2 years) PLUS Lenva 20 mg via oral capsule QD up to at least 2 years. Participants continued study intervention until progressive disease or unacceptable toxicity.
- Cohort D2: Colorectal Cancer (Lenva): Participants received Lenva 24 mg via oral capsule QD up to at least 2 years. Participants continued study intervention until progressive disease or unacceptable toxicity.
Period: Overall Study
Arm/Group | Cohort A: Triple Negative Breast Cancer (Lenva + Pembro) | Cohort B: Ovarian Cancer (Lenva + Pembro) | Cohort C: Gastric Cancer (Lenva + Pembro) | Cohort D1: Colorectal Cancer (Lenva + Pembro) | Cohort D2: Colorectal Cancer (Lenva) | Cohort E: Glioblastoma Multiforma (Lenva + Pembro) | Cohort F: Biliary Tract Cancer (Lenva + Pembro) | Cohort G: Pancreatic Cancer (Lenva + Pembro)
Started | 31 | 31 | 102 | 107 | 32 | 102 | 103 | 103
Treated | 31 | 31 | 99 | 105 | 30 | 101 | 102 | 103
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 31 | 31 | 102 | 107 | 32 | 102 | 103 | 103
Not completed — Lost to Follow-up | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 3 | 0 | 2 | 2 | 3
Not completed — Sponsor Decision | 3 | 3 | 3 | 6 | 0 | 3 | 3 | 2
Not completed — Death | 27 | 28 | 95 | 95 | 30 | 96 | 97 | 98
Not completed — Enrolled in error | 0 | 0 | 3 | 2 | 2 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A: Triple Negative Breast Cancer (Lenva + Pembro) | Cohort B: Ovarian Cancer (Lenva + Pembro) | Cohort C: Gastric Cancer (Lenva + Pembro) | Cohort D1: Colorectal Cancer (Lenva + Pembro) | Cohort D2: Colorectal Cancer (Lenva) | Cohort E: Glioblastoma Multiforma (Lenva + Pembro) | Cohort F: Biliary Tract Cancer (Lenva + Pembro) | Cohort G: Pancreatic Cancer (Lenva + Pembro) | Total
Number analyzed (Participants) | 31 | 31 | 102 | 107 | 32 | 102 | 103 | 103 | 611
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 25 | 18 | 68 | 71 | 25 | 83 | 52 | 56 | 398
  >=65 years | 6 | 13 | 34 | 36 | 7 | 19 | 51 | 47 | 213
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 31 | 30 | 32 | 14 | 38 | 53 | 42 | 271
  Male | 0 | 0 | 72 | 75 | 18 | 64 | 50 | 61 | 340
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 2 | 17 | 19 | 9 | 13 | 9 | 16 | 91
  Not Hispanic or Latino | 19 | 23 | 64 | 77 | 23 | 73 | 76 | 86 | 441
  Unknown or Not Reported | 6 | 6 | 21 | 11 | 0 | 16 | 18 | 1 | 79
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 5 | 4 | 11 | 17 | 2 | 17 | 18 | 8 | 82
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Black or African American | 0 | 0 | 2 | 4 | 2 | 0 | 1 | 2 | 11
  White | 22 | 23 | 70 | 71 | 25 | 72 | 71 | 90 | 444
  More than one race | 0 | 0 | 2 | 4 | 3 | 1 | 0 | 3 | 13
  Unknown or Not Reported | 4 | 4 | 17 | 11 | 0 | 11 | 13 | 0 | 60

OUTCOME MEASURES:

1. Secondary Outcome: Disease Control Rate (DCR) Per RECIST 1.1 by Investigator Assessment
Description: DCR was defined per RECIST 1.1 as the percentage of participants who have a Complete Response (CR: Disappearance of all target lesions) or Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) or Stable Disease (SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease [PD: At least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD]). Disease Control rate per RECIST 1.1 by investigator assessment is presented. Per protocol, only data for Cohorts A and B were presented for this endpoint.
Time Frame: Up to approximately 66 months
Population: All allocated participants who received at least 1 dose of study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A: Triple Negative Breast Cancer (Lenva + Pembro) | Cohort B: Ovarian Cancer (Lenva + Pembro)
Number analyzed (Participants) | 31 | 31
Percentage of Participants | 51.6 [33.1 to 69.8] | 77.4 [58.9 to 90.4]

2. Secondary Outcome: Disease Control Rate (DCR) Per RECIST 1.1 or RANO Criteria (GBM Only) by BICR
Description: DCR was defined per RECIST 1.1 as the percentage of participants who have a Complete Response (CR: Disappearance of all target lesions) or Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) or Stable Disease (SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease [PD: At least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm]). The appearance of one or more new lesions is also considered PD.]). For participants with GBM, response was assessed according to RANO criteria whereby overall response was based on both radiographic response (CR: disappearance of all target lesions, PR: sum of products of diameters [SPD] decreased by ≥ 50% from baseline value and SD: SPD <50% decreased from baseline, but <25% increased from nadir) and clinical performance status with steroid dose information. The DCR as assessed by BICR is presented.
Time Frame: Up to approximately 66 months
Population: All allocated participants who received at least 1 dose of study intervention. Per protocol, only data for Cohorts C, D1, D2, E, F, and G were presented for this endpoint.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort C: Gastric Cancer (Lenva + Pembro) | Cohort D1: Colorectal Cancer (Lenva + Pembro) | Cohort D2: Colorectal Cancer (Lenva) | Cohort E: Glioblastoma Multiforma (Lenva + Pembro) | Cohort F: Biliary Tract Cancer (Lenva + Pembro) | Cohort G: Pancreatic Cancer (Lenva + Pembro)
Number analyzed (Participants) | 99 | 105 | 30 | 101 | 102 | 103
Percentage of Participants | 53.5 [43.2 to 63.6] | 52.4 [42.4 to 62.2] | 56.7 [37.4 to 74.5] | 57.4 [47.2 to 67.2] | 64.7 [54.6 to 73.9] | 37.9 [28.5 to 48.0]

3. Secondary Outcome: Duration of Response (DOR) Per RECIST 1.1 by Investigator Assessment
Description: For participants who demonstrate a confirmed Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1, DOR was defined as the time from first documented evidence of CR or PR until progressive disease (PD) or death. Per RECIST 1.1, PD is defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD. Duration of response per RECIST 1.1 by investigator assessment is presented. Per protocol, only data for Cohorts A and B were presented for this endpoint.
Time Frame: Up to approximately 66 months
Population: All allocated participants who received at least 1 dose of study intervention and had confirmed complete response or partial response.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort A: Triple Negative Breast Cancer (Lenva + Pembro) | Cohort B: Ovarian Cancer (Lenva + Pembro)
Number analyzed (Participants) | 7 | 8
Months | 22.9 [4.2 to NA] — NA = Upper limit not reached at time of data cut-off due to insufficient number of responding participants with relapse. | 15.3 [6.4 to NA] — NA = Upper limit not reached at time of data cut-off due to insufficient number of responding participants with relapse.

4. Secondary Outcome: Duration of Response (DOR) Per RECIST 1.1 or RANO Criteria (GBM Only) by BICR
Description: For participants who demonstrate a confirmed Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1, DOR was defined as the time from first documented evidence of CR or PR until progressive disease (PD) or death. Per RECIST 1.1, PD is defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD. For participants with GBM, response will be assessed according to RANO criteria whereby overall RANO response is based on both radiographic response (CR: disappearance of all target lesions, PR: SPD decreased by ≥ 50% from baseline value) and clinical performance status with steroid dose information. DOR assessments were based on blinded central imaging review with confirmation.
Time Frame: Up to approximately 66 months
Population: All allocated participants who received at least 1 dose of study intervention and had confirmed complete response or partial response. Per protocol, only data for Cohorts C, D1, D2, E, F, and G were presented for this endpoint.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort C: Gastric Cancer (Lenva + Pembro) | Cohort D1: Colorectal Cancer (Lenva + Pembro) | Cohort D2: Colorectal Cancer (Lenva) | Cohort E: Glioblastoma Multiforma (Lenva + Pembro) | Cohort F: Biliary Tract Cancer (Lenva + Pembro) | Cohort G: Pancreatic Cancer (Lenva + Pembro)
Number analyzed (Participants) | 15 | 15 | 2 | 22 | 18 | 8
Months | 8.3 [4.2 to NA] — NA = Upper limit not reached at time of data cut-off due to insufficient number of responding participants with relapse. | 8.3 [4.2 to 18.5] | NA [NA to NA] — NA = Median, Lower and Upper limit not reached at time of data cut-off due to insufficient number of responding participants with relapse. | 4.6 [3.2 to 15.6] | 6.2 [4.2 to 7.1] | 5.8 [2.7 to NA] — NA = Upper limit not reached at time of data cut-off due to insufficient number of responding participants with relapse.

5. Secondary Outcome: Progression-Free Survival (PFS) Per RECIST 1.1 by Investigator Assessment
Description: PFS was defined as the time from date of study treatment to the first documented progressive disease (PD) based on RECIST 1.1, modified to follow a maximum of 10 target lesions and a maximum of 5 target lesions per organ or death due to any cause, whichever occurred first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD. The percentage of participants who experienced PFS per RECIST 1.1 by investigator assessment is presented. Per protocol, only data for Cohorts A and B were presented for this endpoint.
Time Frame: Up to approximately 66 months
Population: All allocated participants who received at least 1 dose of study intervention.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort A: Triple Negative Breast Cancer (Lenva + Pembro) | Cohort B: Ovarian Cancer (Lenva + Pembro)
Number analyzed (Participants) | 31 | 31
Months | 4.2 [1.7 to 6.3] | 6.1 [4.1 to 9.4]

6. Secondary Outcome: Progression-Free Survival (PFS) Per RECIST 1.1 or RANO Criteria (GBM Only) by BICR
Description: PFS was defined as the time from date of study treatment to the first documented progressive disease (PD) based on RECIST 1.1 (or RANO for GBM participants), modified to follow a maximum of 10 target lesions and a maximum of 5 target lesions per organ or death due to any cause, whichever occurred first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD. For participants with GBM, either radiological progression or clinical deterioration (not attributable to a nontumor-related cause) qualifies as PD. The percentage of participants who experienced PFS per RECIST 1.1 or RANO by BICR is presented. Per protocol, only data for Cohorts C, D1, D2, E, F, and G were presented for this endpoint.
Time Frame: Up to approximately 66 months
Population: All allocated participants who received at least 1 dose of study intervention.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort C: Gastric Cancer (Lenva + Pembro) | Cohort D1: Colorectal Cancer (Lenva + Pembro) | Cohort D2: Colorectal Cancer (Lenva) | Cohort E: Glioblastoma Multiforma (Lenva + Pembro) | Cohort F: Biliary Tract Cancer (Lenva + Pembro) | Cohort G: Pancreatic Cancer (Lenva + Pembro)
Number analyzed (Participants) | 99 | 105 | 30 | 101 | 102 | 103
Months | 3.5 [2.3 to 4.1] | 3.4 [2.1 to 4.1] | 3.4 [2.1 to 4.8] | 3.0 [2.8 to 4.1] | 4.1 [3.6 to 5.9] | 2.1 [2.1 to 3.1]

7. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of study treatment to the date of death due to any cause. Participants without documented death at the time of the final analysis were censored at the date of the last follow-up. The OS for all participants is presented.
Time Frame: Up to approximately 66 months
Population: All allocated participants who received at least 1 dose of study intervention.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort A: Triple Negative Breast Cancer (Lenva + Pembro) | Cohort B: Ovarian Cancer (Lenva + Pembro) | Cohort C: Gastric Cancer (Lenva + Pembro) | Cohort D1: Colorectal Cancer (Lenva + Pembro) | Cohort D2: Colorectal Cancer (Lenva) | Cohort E: Glioblastoma Multiforma (Lenva + Pembro) | Cohort F: Biliary Tract Cancer (Lenva + Pembro) | Cohort G: Pancreatic Cancer (Lenva + Pembro)
Number analyzed (Participants) | 31 | 31 | 99 | 105 | 30 | 101 | 102 | 103
Months | 11.4 [4.1 to 21.7] | 21.3 [11.7 to 32.3] | 4.7 [3.8 to 6.1] | 8.7 [7.0 to 10.0] | 7.9 [5.6 to 14.9] | 8.6 [7.4 to 10.8] | 7.9 [5.6 to 9.5] | 4.3 [3.8 to 5.4]

8. Secondary Outcome: Area Under the Concentration Curve at Steady State (AUCss) of Lenvatinib
Description: Blood samples were collected at pre-specified timepoints to determine the AUCss in participants receiving Lenvatinib (Lenva) co-administered with Pembrolizumab (Pembro). AUCss was defined as a measure of drug exposure that was calculated as the product of plasma drug concentration and time after drug administration at steady state. AUCss determined by blood samples collected pre-dose and at designated timepoints post-dose are presented. Noncompartmental analysis was used to calculate AUC0ss for each participant. Mean and standard deviation of AUCss were calculated for each cohort. As specified in the protocol, pharmacokinetic analysis was not planned or conducted in Cohorts D2 and G.
Time Frame: Cycle 1 Day 1: 0.5-4 hours and 6-10 hours post-dose; Cycle 1 Day 15: pre-dose and 2-12 hours post-dose; Cycle 2 Day 1: pre-dose, 0.5-4 hours, and 6-10 hours post-dose (up to approximately 23 days). Each cycle is 21 days.
Population: All allocated participants who received at least 1 dose of study intervention and had data available for this endpoint.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Cohort A: Triple Negative Breast Cancer (Lenva + Pembro) | Cohort B: Ovarian Cancer (Lenva + Pembro) | Cohort C: Gastric Cancer (Lenva + Pembro) | Cohort D1: Colorectal Cancer (Lenva + Pembro) | Cohort E: Glioblastoma Multiforma (Lenva + Pembro) | Cohort F: Biliary Tract Cancer (Lenva + Pembro)
Number analyzed (Participants) | 30 | 31 | 93 | 104 | 100 | 100
ng*hr/mL | 3253 (1029) | 3145 (984) | 2392 (803) | 2994 (1143) | 2617 (804) | 2886 (838)

9. Primary Outcome: Objective Response Rate (ORR) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) by Investigator Assessment
Description: ORR was defined as the percentage of participants who had a best overall response of either Complete Response (CR): Disappearance of all target lesions or Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions as assessed by RECIST 1.1. The percentage of participants who experienced a CR or PR as assessed by RECIST 1.1 by investigator assessment was presented. Per protocol, only data for Cohorts A and B were presented for this endpoint.
Time Frame: Up to approximately 66 months
Population: All allocated participants who received at least 1 dose of study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A: Triple Negative Breast Cancer (Lenva + Pembro) | Cohort B: Ovarian Cancer (Lenva + Pembro)
Number analyzed (Participants) | 31 | 31
Percentage of Participants | 22.6 [9.6 to 41.1] | 25.8 [11.9 to 44.6]

10. Primary Outcome: Objective Response Rate (ORR) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) or Response Assessment in Neuro-Oncology (RANO) Criteria (for Glioblastoma Multiforma [GBM] Only), by Blinded Independent Central Review (BICR)
Description: ORR was defined as the percentage of participants who had a best overall response of either Complete Response (CR): Disappearance of all target lesions or Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions as assessed by RECIST 1.1. For participants with GBM, response was assessed according to RANO criteria whereby ORR was defined as the percentage of participants who had a best overall response of either Complete response (CR): Disappearance of all target lesions or Partial response (PR): sum of products of diameters decreased by ≥50% from baseline value. The percentage of participants who experienced a CR or PR as assessed by RECIST 1.1 or RANO by BICR was presented. Per protocol, only data for Cohorts C, D1, D2, E, F, and G were presented for this endpoint.
Time Frame: Up to approximately 66 months
Population: All allocated participants who received at least 1 dose of study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Cohort C: Gastric Cancer (Lenva + Pembro): Participants received Pembro 200 mg via IV infusion on Day 1 of each 21-day cycle (Q3W) for up to 35 cycles (up to 2 years) PLUS Lenva 20 mg via oral capsule once a day (QD) up to at least 2 years. Participants continued study intervention until progressive disease or unacceptable toxicity.
Arm/Group | Cohort C: Gastric Cancer (Lenva + Pembro) | Cohort D1: Colorectal Cancer (Lenva + Pembro) | Cohort D2: Colorectal Cancer (Lenva) | Cohort E: Glioblastoma Multiforma (Lenva + Pembro) | Cohort F: Biliary Tract Cancer (Lenva + Pembro) | Cohort G: Pancreatic Cancer (Lenva + Pembro)
Number analyzed (Participants) | 99 | 105 | 30 | 101 | 102 | 103
Percentage of Participants | 15.2 [8.7 to 23.8] | 14.3 [8.2 to 22.5] | 6.7 [0.8 to 22.1] | 21.8 [14.2 to 31.1] | 17.6 [10.8 to 26.4] | 7.8 [3.4 to 14.7]

11. Primary Outcome: Number of Participants With One or More Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants with at least one or more AE is presented.
Time Frame: Up to approximately 66 months
Population: All allocated participants who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Triple Negative Breast Cancer (Lenva + Pembro) | Cohort B: Ovarian Cancer (Lenva + Pembro) | Cohort C: Gastric Cancer (Lenva + Pembro) | Cohort D1: Colorectal Cancer (Lenva + Pembro) | Cohort D2: Colorectal Cancer (Lenva) | Cohort E: Glioblastoma Multiforma (Lenva + Pembro) | Cohort F: Biliary Tract Cancer (Lenva + Pembro) | Cohort G: Pancreatic Cancer (Lenva + Pembro)
Number analyzed (Participants) | 31 | 31 | 99 | 105 | 30 | 101 | 102 | 103
Participants | 31 | 31 | 97 | 104 | 30 | 101 | 102 | 103

12. Primary Outcome: Number of Participants Who Discontinued From Study Treatment Due to an AE
Description: An AE was defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants who discontinued from study treatment due to an AE is presented.
Time Frame: Up to approximately 62 months
Population: All allocated participants who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Triple Negative Breast Cancer (Lenva + Pembro) | Cohort B: Ovarian Cancer (Lenva + Pembro) | Cohort C: Gastric Cancer (Lenva + Pembro) | Cohort D1: Colorectal Cancer (Lenva + Pembro) | Cohort D2: Colorectal Cancer (Lenva) | Cohort E: Glioblastoma Multiforma (Lenva + Pembro) | Cohort F: Biliary Tract Cancer (Lenva + Pembro) | Cohort G: Pancreatic Cancer (Lenva + Pembro)
Number analyzed (Participants) | 31 | 31 | 99 | 105 | 30 | 101 | 102 | 103
Participants | 5 | 11 | 23 | 19 | 4 | 11 | 20 | 19

ADVERSE EVENTS:
Time Frame: Up to approximately 66 months
Description: All-Cause Mortality included all randomized participants. Serious and Other adverse events (AEs) included all randomized participants who received at least one dose of study intervention. Per protocol, disease progression of cancer on study was not considered an AE unless considered related to study intervention. MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" and "Disease progression" not related to study intervention were excluded.
Arm/Group | Cohort A: Triple Negative Breast Cancer (Lenva + Pembro) | Cohort B: Ovarian Cancer (Lenva + Pembro) | Cohort C: Gastric Cancer (Lenva + Pembro) | Cohort D1: Colorectal Cancer (Lenva + Pembro) | Cohort D2: Colorectal Cancer (Lenva) | Cohort E: Glioblastoma Multiforma (Lenva + Pembro) | Cohort F: Biliary Tract Cancer (Lenva + Pembro) | Cohort G: Pancreatic Cancer (Lenva + Pembro)
All-Cause Mortality (participants affected / at risk) | 27/31 | 28/31 | 97/102 | 97/107 | 30/32 | 99/102 | 98/103 | 101/103
Serious Adverse Events (participants affected / at risk) | 16/31 | 19/31 | 57/99 | 55/105 | 12/30 | 30/101 | 62/102 | 49/103
Other Adverse Events (participants affected / at risk) | 30/31 | 31/31 | 95/99 | 103/105 | 29/30 | 98/101 | 100/102 | 101/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A: Triple Negative Breast Cancer (Lenva + Pembro) (N=31) | Cohort B: Ovarian Cancer (Lenva + Pembro) (N=31) | Cohort C: Gastric Cancer (Lenva + Pembro) (N=99) | Cohort D1: Colorectal Cancer (Lenva + Pembro) (N=105) | Cohort D2: Colorectal Cancer (Lenva) (N=30) | Cohort E: Glioblastoma Multiforma (Lenva + Pembro) (N=101) | Cohort F: Biliary Tract Cancer (Lenva + Pembro) (N=102) | Cohort G: Pancreatic Cancer (Lenva + Pembro) (N=103)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity myocarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypophysitis (Endocrine disorders) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 4 (4) | 2 (3) | 0 (0) | 0 (0) | 6 (8) | 5 (6)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal wall haematoma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 3 (3) | 3 (4) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Duodenal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Duodenal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Duodenal stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Immune-mediated pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal dilatation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Intestinal pseudo-obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Jejunal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Obstruction gastric (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Varices oesophageal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 4 (4) | 7 (9) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Biliary obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 5 (5) | 1 (1)
Biliary tract disorder (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 6 (6) | 0 (0)
Cholangitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Jaundice (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal wall abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anorectal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Bacteroides infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Biliary sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Biliary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Device related sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Encephalitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Escherichia sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Extradural abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infective aneurysm (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Liver abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meningitis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Periorbital cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2) | 2 (3) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Scrotal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vascular device infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal anastomosis complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stomal hernia (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract stoma complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Embolic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intracranial pressure increased (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Leukoencephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myasthenic syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neurotoxicity (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paraneoplastic neurological syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal cord compression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal cord haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Status epilepticus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Vascular encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vasogenic cerebral oedema (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wernicke's encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device dislocation (Product Issues) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stent malfunction (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disorientation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (2) | 4 (4) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nephrotic syndrome (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Loss of personal independence in daily activities (Social circumstances) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Assisted suicide (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertensive urgency (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iliac artery occlusion (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vasculitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Venous haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A: Triple Negative Breast Cancer (Lenva + Pembro) (N=31) | Cohort B: Ovarian Cancer (Lenva + Pembro) (N=31) | Cohort C: Gastric Cancer (Lenva + Pembro) (N=99) | Cohort D1: Colorectal Cancer (Lenva + Pembro) (N=105) | Cohort D2: Colorectal Cancer (Lenva) (N=30) | Cohort E: Glioblastoma Multiforma (Lenva + Pembro) (N=101) | Cohort F: Biliary Tract Cancer (Lenva + Pembro) (N=102) | Cohort G: Pancreatic Cancer (Lenva + Pembro) (N=103)
Anaemia (Blood and lymphatic system disorders) | 5 (9) | 4 (5) | 17 (20) | 12 (19) | 6 (8) | 3 (8) | 11 (13) | 15 (17)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 5 (5) | 2 (2) | 0 (0) | 2 (3) | 1 (1) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 2 (3) | 6 (7) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 4 (5)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 2 (3) | 10 (14) | 9 (10) | 3 (3) | 7 (8) | 4 (5) | 10 (13)
Tachycardia (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 4 (4) | 2 (2) | 6 (6) | 9 (9) | 1 (1) | 6 (8) | 6 (6) | 3 (3)
Hypothyroidism (Endocrine disorders) | 14 (15) | 14 (14) | 25 (25) | 46 (53) | 12 (13) | 28 (30) | 34 (35) | 28 (29)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 5 (6) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 4 (4) | 5 (6)
Abdominal pain (Gastrointestinal disorders) | 5 (7) | 10 (11) | 17 (19) | 25 (28) | 5 (7) | 12 (14) | 32 (44) | 29 (34)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 8 (10) | 7 (7) | 8 (9) | 2 (2) | 4 (4) | 10 (10) | 7 (8)
Ascites (Gastrointestinal disorders) | 0 (0) | 4 (5) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 6 (6) | 4 (4)
Constipation (Gastrointestinal disorders) | 7 (7) | 11 (11) | 17 (18) | 22 (25) | 3 (3) | 14 (15) | 24 (27) | 19 (24)
Diarrhoea (Gastrointestinal disorders) | 14 (34) | 19 (38) | 30 (40) | 47 (74) | 16 (44) | 26 (43) | 42 (67) | 25 (41)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 8 (9) | 2 (2) | 7 (9) | 1 (1) | 4 (4) | 11 (11) | 8 (9)
Dyspepsia (Gastrointestinal disorders) | 5 (6) | 2 (3) | 4 (4) | 9 (9) | 0 (0) | 3 (3) | 8 (9) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 6 (6) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 3 (3)
Flatulence (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 3 (4)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (4) | 3 (4) | 4 (4) | 5 (5) | 1 (1) | 2 (2) | 3 (3) | 2 (2)
Nausea (Gastrointestinal disorders) | 13 (17) | 15 (21) | 31 (32) | 34 (45) | 5 (7) | 19 (21) | 37 (55) | 37 (50)
Stomatitis (Gastrointestinal disorders) | 4 (4) | 6 (6) | 9 (9) | 12 (13) | 4 (5) | 6 (6) | 12 (15) | 9 (9)
Toothache (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 3 (3) | 3 (3)
Vomiting (Gastrointestinal disorders) | 10 (18) | 13 (22) | 15 (17) | 26 (34) | 8 (11) | 13 (13) | 20 (43) | 19 (26)
Asthenia (General disorders) | 7 (8) | 6 (8) | 30 (34) | 27 (35) | 7 (8) | 29 (36) | 23 (29) | 23 (25)
Chest pain (General disorders) | 3 (3) | 1 (1) | 5 (5) | 2 (2) | 1 (1) | 3 (3) | 4 (4) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 6 (6) | 6 (6)
Fatigue (General disorders) | 13 (14) | 14 (16) | 21 (22) | 41 (47) | 9 (11) | 20 (22) | 40 (52) | 31 (35)
Influenza like illness (General disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 7 (10) | 10 (10) | 9 (10) | 10 (12) | 2 (2) | 11 (14) | 15 (18) | 5 (5)
Oedema peripheral (General disorders) | 2 (3) | 5 (5) | 5 (5) | 15 (16) | 0 (0) | 5 (5) | 13 (13) | 19 (20)
Peripheral swelling (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 4 (4) | 3 (3) | 8 (9) | 11 (14) | 2 (2) | 8 (13) | 11 (15) | 19 (23)
Cystitis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gingivitis (Infections and infestations) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Tooth infection (Infections and infestations) | 0 (0) | 2 (3) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (3) | 5 (10) | 4 (4) | 7 (8) | 3 (5) | 6 (8) | 7 (7) | 5 (5)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 9 (9) | 0 (0) | 3 (3)
Alanine aminotransferase increased (Investigations) | 5 (12) | 7 (17) | 12 (18) | 24 (34) | 10 (14) | 22 (33) | 21 (25) | 14 (17)
Amylase increased (Investigations) | 1 (1) | 2 (2) | 7 (9) | 7 (10) | 3 (3) | 6 (10) | 3 (4) | 6 (8)
Aspartate aminotransferase increased (Investigations) | 6 (11) | 8 (17) | 18 (25) | 24 (35) | 7 (8) | 20 (27) | 26 (31) | 19 (24)
Blood albumin decreased (Investigations) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 2 (2)
Blood alkaline phosphatase increased (Investigations) | 2 (2) | 6 (7) | 14 (14) | 13 (15) | 11 (14) | 4 (4) | 14 (14) | 9 (13)
Blood bilirubin increased (Investigations) | 1 (3) | 2 (2) | 7 (8) | 15 (24) | 6 (8) | 7 (7) | 15 (17) | 8 (9)
Blood cholesterol increased (Investigations) | 1 (4) | 0 (0) | 0 (0) | 6 (12) | 1 (1) | 6 (6) | 1 (1) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 3 (3) | 0 (0) | 1 (2) | 2 (4)
Blood creatinine increased (Investigations) | 1 (1) | 1 (1) | 5 (7) | 12 (17) | 3 (6) | 3 (3) | 6 (8) | 11 (11)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 1 (1) | 4 (4) | 3 (3) | 2 (2) | 5 (9) | 0 (0) | 4 (4)
Blood magnesium decreased (Investigations) | 1 (1) | 1 (1) | 2 (4) | 1 (1) | 3 (4) | 0 (0) | 1 (1) | 0 (0)
Blood sodium increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 1 (6) | 3 (3) | 3 (3) | 8 (17) | 4 (5) | 7 (11) | 3 (3) | 3 (3)
Blood urea increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 2 (2) | 1 (1) | 0 (0) | 3 (4)
Gamma-glutamyltransferase increased (Investigations) | 2 (2) | 2 (2) | 7 (7) | 3 (4) | 1 (1) | 3 (3) | 4 (4) | 1 (1)
Lipase increased (Investigations) | 2 (2) | 3 (4) | 8 (9) | 12 (14) | 3 (3) | 5 (5) | 6 (8) | 7 (10)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 4 (5) | 2 (2) | 7 (11) | 4 (5) | 2 (3)
Neutrophil count decreased (Investigations) | 5 (10) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 1 (1) | 5 (6)
Platelet count decreased (Investigations) | 5 (7) | 3 (3) | 9 (10) | 8 (10) | 6 (8) | 7 (8) | 7 (7) | 12 (17)
Platelet count increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 3 (5) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Protein total decreased (Investigations) | 1 (1) | 0 (0) | 3 (4) | 3 (5) | 2 (3) | 4 (9) | 1 (1) | 4 (7)
Weight decreased (Investigations) | 8 (9) | 7 (8) | 15 (15) | 13 (13) | 8 (9) | 6 (6) | 10 (10) | 22 (23)
Decreased appetite (Metabolism and nutrition disorders) | 9 (12) | 15 (20) | 30 (31) | 46 (50) | 6 (6) | 19 (20) | 37 (44) | 33 (40)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 4 (5) | 0 (0) | 1 (1) | 2 (3) | 2 (2) | 2 (2) | 4 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (6) | 1 (3) | 3 (3) | 6 (7) | 3 (4) | 5 (11) | 3 (3) | 7 (9)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 4 (5) | 4 (4) | 3 (5) | 1 (1) | 1 (4) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (4) | 0 (0) | 1 (1) | 6 (17) | 1 (2) | 2 (5) | 1 (1) | 2 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (2) | 4 (5) | 9 (9) | 11 (11) | 5 (5) | 2 (3) | 6 (7) | 9 (11)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (4) | 3 (6) | 4 (4) | 4 (7) | 2 (2) | 9 (11) | 8 (12) | 13 (15)
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 (5) | 5 (17) | 1 (1) | 5 (6) | 6 (9) | 5 (9) | 7 (9) | 4 (5)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 8 (8) | 5 (6) | 1 (1) | 2 (3) | 12 (14) | 12 (15)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 5 (5) | 5 (5) | 2 (2) | 4 (4) | 3 (4) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 (18) | 11 (17) | 10 (13) | 21 (26) | 4 (4) | 12 (15) | 18 (22) | 16 (19)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 4 (4) | 13 (14) | 20 (23) | 1 (1) | 4 (4) | 15 (15) | 12 (12)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (4) | 1 (1) | 4 (4) | 1 (1) | 3 (3) | 3 (3) | 3 (3)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 2 (2) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 6 (6) | 1 (1) | 0 (0) | 4 (4) | 3 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 7 (7) | 6 (6) | 17 (17) | 3 (3) | 8 (8) | 6 (7) | 5 (5)
Neck pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 3 (3) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 4 (6) | 6 (8) | 2 (2) | 6 (7) | 5 (6) | 1 (2)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 8 (8) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 5 (5) | 4 (4) | 7 (7) | 0 (0) | 4 (4) | 3 (4) | 5 (5)
Dysgeusia (Nervous system disorders) | 2 (2) | 4 (5) | 5 (5) | 2 (2) | 1 (1) | 4 (4) | 5 (5) | 9 (9)
Headache (Nervous system disorders) | 10 (16) | 10 (16) | 7 (8) | 18 (21) | 6 (11) | 25 (29) | 25 (28) | 22 (25)
Tremor (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 2 (2) | 3 (3)
Anxiety (Psychiatric disorders) | 2 (2) | 5 (6) | 2 (2) | 9 (9) | 0 (0) | 5 (6) | 1 (1) | 2 (2)
Depression (Psychiatric disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 4 (4) | 2 (2) | 4 (4)
Insomnia (Psychiatric disorders) | 3 (3) | 1 (1) | 5 (5) | 9 (10) | 0 (0) | 5 (5) | 6 (6) | 8 (10)
Dysuria (Renal and urinary disorders) | 0 (0) | 3 (3) | 2 (2) | 3 (3) | 1 (1) | 6 (6) | 1 (1) | 3 (4)
Haematuria (Renal and urinary disorders) | 1 (1) | 2 (2) | 3 (3) | 4 (4) | 2 (2) | 4 (5) | 2 (2) | 2 (2)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Leukocyturia (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 6 (8) | 13 (18) | 12 (13) | 39 (52) | 11 (12) | 12 (15) | 23 (24) | 22 (25)
Breast pain (Reproductive system and breast disorders) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 4 (5) | 6 (6) | 10 (10) | 1 (1) | 9 (9) | 11 (15) | 5 (5)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3) | 20 (20) | 21 (21) | 12 (14) | 11 (12) | 31 (34) | 17 (18)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (5) | 6 (6) | 7 (8) | 2 (2) | 5 (5) | 14 (15) | 7 (8)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 8 (8) | 4 (4) | 0 (0) | 5 (6) | 9 (11) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 3 (3) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 6 (6) | 6 (6) | 1 (1) | 4 (4) | 7 (7) | 7 (7)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 8 (8) | 6 (6) | 10 (10) | 8 (8) | 5 (6) | 10 (10) | 12 (13) | 12 (14)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (3) | 6 (7) | 13 (13) | 9 (10) | 0 (0) | 4 (4) | 15 (20) | 8 (11)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 5 (5) | 4 (4) | 13 (16) | 2 (3) | 14 (18) | 16 (19) | 15 (17)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 5 (5) | 0 (0) | 1 (1) | 4 (5) | 4 (4)
Hypertension (Vascular disorders) | 16 (25) | 21 (28) | 37 (42) | 59 (92) | 17 (22) | 51 (65) | 58 (74) | 55 (65)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (4) | 1 (1) | 0 (0) | 6 (7) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor will generally support publication of multicenter studies only in their entirety and not as individual site data. In this case, a coordinating investigator will be designated by mutual agreement. If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. Authorship will be determined by mutual agreement and in line with ICMJE authorship requirements.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-18): https://cdn.clinicaltrials.gov/large-docs/26/NCT03797326/Prot_SAP_000.pdf